CLINICAL TRIAL: NCT03148795
Title: TALAPRO-1: A PHASE 2, OPEN-LABEL, RESPONSE RATE STUDY OF TALAZOPARIB IN MEN WITH DNA REPAIR DEFECTS AND METASTATIC CASTRATION-RESISTANT PROSTATE CANCER WHO PREVIOUSLY RECEIVED TAXANE-BASED CHEMOTHERAPY AND PROGRESSED ON AT LEAST 1 NOVEL HORMONAL AGENT (ENZALUTAMIDE AND/OR ABIRATERONE ACETATE/PREDNISONE)
Brief Title: A Study of Talazoparib in Men With DNA Repair Defects and Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDV3800-06; C3441006 (Other: Alias Study Number); 2016-002036-32 (EudraCT Number)
Record Dates: First submitted 2017-05-09; First posted 2017-05-11 (Actual); Results first posted 2021-09-08 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — talazoparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Talazoparib (Experimental): Talazoparib 1 mg daily
  Interventions: Drug: Talazoparib

INTERVENTIONS:
Drug: Talazoparib — 1 mg daily
  Other Names: MDV3800

SUMMARY:
The purpose of this international, phase 2, open-label, response rate study of talazoparib is to assess the efficacy and safety of talazoparib in men with DNA repair defects metastatic castration-resistant prostate cancer (CRPC) who previously received taxane-based chemotherapy and progressed on at least 1 novel hormonal agent (enzalutamide and/or abiraterone acetate/prednisone).

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Histologically or cytologically confirmed adenocarcinoma of the prostate without signet cell, or small cell features.
3. Patients must have measurable soft tissue disease per RECIST 1.1
4. DNA damage repair deficiency as assessed centrally by a gene mutation biomarker panel (testing of de novo or archival tumor tissue (via central laboratory) or prior historical testing (with Sponsor approval) using the Foundation Medicine, FoundationOne CDx™ NGS gene panel test.
5. Consent to a saliva sample collection for a germline comparator, unless prohibited by local regulations or ethics committee (EC) decision.
6. Serum testosterone ≤ 1.73 nmol/L (50 ng/dL) at screening.
7. Bilateral orchiectomy or ongoing androgen deprivation therapy with a gonadotropin-releasing hormone (GnRH) agonist/antagonist (surgical or medical castration).
8. Progressive disease at study entry defined as 1 or more of the following 3 criteria:

   * A minimum of 3 rising PSA values with an interval of at least 1 week between determinations. The screening central laboratory PSA value must be ≥ 2 μg/L (2 ng/mL) if qualifying solely by PSA progression.
   * Soft tissue disease progression as defined by RECIST 1.1.
   * Bone disease progression defined by PCWG3 with 2 or more new metastatic lesions on bone scan.
9. Metastatic disease.
10. Previous treatment with 1 or 2 chemotherapy regimens including at least 1 taxane-based regimen for metastatic (non castrate or castrate) prostate cancer. Patients may have received radium-223 and/or cabazitaxel, or were deemed unsuitable, declined, or did not have access to these therapies.
11. Documented disease progression (either radiographic or biochemical) on at least 1 novel hormonal therapy (enzalutamide and/or abiraterone acetate/prednisone) for the treatment of metastatic CRPC, irrespective of prior NHT treatment for non castrate prostate cancer or nonmetastatic (M0) CRPC.
12. Bisphosphonate or denosumab dosage must have been stable for at least 4 weeks before day 1 for patients receiving these therapies.
13. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
14. Estimated life expectancy of ≥ 6 months as assessed by the investigator.
15. Able to swallow the study drug, have no known intolerance to study drugs or excipients, and comply with study requirements.
16. Must use a condom when having sex from the time of the first dose of study drug through 4 months after last dose of study drug. A highly effective form of contraception must be used from the time of the first dose of study drug through 4 months after last dose of study drug when having sex with a non pregnant female partner of childbearing potential.
17. Must agree not to donate sperm from the first dose of study drug to 4 months after the last dose of study drug.
18. Patients must be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

1. 1. Use of systemic chemotherapeutic (including but not limited to taxanes), hormonal, biologic, or radionuclide therapy for treatment of metastatic prostate cancer (other than approved bone targeting agents and GnRH agonist/antagonist) or any other investigational agent within 4 weeks before day 1.
2. Prior treatment with a PARP inhibitor, cyclophosphamide, or mitoxantrone chemotherapy. Patients who discontinued prior platinum based chemotherapy <=6 months prior to screening or whose disease previously progressed on platinum based therapy at any time in the past are also excluded.
3. Treatment with any concurrent cytotoxic chemotherapy or investigational drug(s) within 4 weeks or 5 half lives of the drug (whichever is longer) before Day 1 and/or during study participation
4. Radiation therapy within 3 weeks (within 2 weeks, if single fraction of radiotherapy) before day 1.
5. Major surgery within 2 weeks before day 1.
6. Clinically significant cardiovascular disease.
7. Significant renal, hepatic, or bone marrow organ dysfunction.
8. Known or suspected brain metastasis or active leptomeningeal disease.
9. Symptomatic or impending spinal cord compression or cauda equina syndrome.
10. Prior diagnosis of myelodysplastic syndrome or acute myeloid leukemia
11. History of another cancer within 3 years before enrollment with the exception of nonmelanoma skin cancers, or American Joint Committee on Cancer stage 0 or stage 1 cancer that has a remote probability of recurrence in the opinion of the investigator and the sponsor.
12. Gastrointestinal disorder affecting absorption.
13. Current or anticipated use within 7 days prior to first dose of study drug or anticipated use during the study of the following P gp inhibitors (amiodarone, carvedilol, clarithromycin, cobicistat, darunavir, dronedarone, erythromycin, indinavir, itraconazole, ketoconazole, lapatinib, lopinavir, propafenone, quinidine, ranolazine, ritonavir, saquinavir, telaprevir, tipranavir, verapamil, and valspodar).
14. Any other acute or chronic medical or psychiatric condition (concurrent disease, infection, or comorbidity) that interferes with ability to participate in the study, causes undue risk, or complicates the interpretation of data, in the opinion of the investigator or sponsor, including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
15. Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or patients who are Pfizer employees, including their family members, directly involved in the conduct of the study.
16. Fertile male subjects who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 4 months after the last dose of investigational product.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 128 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (120):
- United States (42):
  - Arizona Oncology Associates, Tempe, Arizona
  - City of Hope (City of Hope National Medical Center, City of Hope Medical Center), Duarte, California
  - City of Hope-Antelope Valley, Lancaster, California
  - UC Irvine Health Investigational Drug Pharmacy, Orange, California
  - University of California, Irvine Medical Center, Orange, California
  - Medical Oncology Associates-SD, San Diego, California
  - Sharp Outpatient Infusion Therapy Center, San Diego, California
  - Sharp Rees-Stealy, San Diego, California
  - Emory University Hospital, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Piedmont Cancer Institute, PC, Fayetteville, Georgia
  - Piedmont Cancer Institute, PC, Newnan, Georgia
  - Siteman Cancer Center - St. Peters, City of Saint Peters, Missouri
  - Siteman Cancer Center - West County, Creve Coeur, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center - South County, St Louis, Missouri
  - Christian Hospital North East, St Louis, Missouri
  - Weill Cornell Medical Center - New York Presbyterian Hospital, New York, New York
  - Weill Cornell Medical Center-New York Presbyterian Hospital, New York, New York
  - Levine Cancer Institute-Albermarle, Albemarle, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Levine Cancer Institute-Pineville, Charlotte, North Carolina
  - Levine Cancer Institute-Southpark, Charlotte, North Carolina
  - Levine Cancer Institute-University, Charlotte, North Carolina
  - Levine Cancer Institute-Ballantyne, Charlotte, North Carolina
  - Levine Cancer Institute- Gaston, Gastonia, North Carolina
  - Levine Cancer Institute-Lincolnton, Lincolnton, North Carolina
  - Levine Cancer Institute-Monroe, Monroe, North Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Parkway Surgery Center, Myrtle Beach, South Carolina
  - Levine Cancer Institute-Rock Hill, Rock Hill, South Carolina
  - The University of Texas Health Science Center at Tyler dba UT Health East Texas HOPE Cancer Center, Tyler, Texas
  - Virginia Oncology Associates, Hampton, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Swedish Cancer Institute Edmonds Campus, Edmonds, Washington
  - Swedish Cancer Institute Issaquah Campus, Issaquah, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
  - Froedtert Hospital/Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (16):
  - Medical Imaging St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - St Vincent's Hospital Sydney, The Kinghorn Cancer Centre, Darlinghurst, New South Wales
  - PRP Diagnostic Imaging, Westmead, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Icon Cancer Care Wesley, Auchenflower, Queensland
  - Liz Plummer Cancer Care Center, Cairns, Queensland
  - Icon Cancer Care Chermside, Chermside, Queensland
  - Icon Cancer Care South Brisbane, South Brisbane, Queensland
  - Icon Cancer Care, South Brisbane, Queensland
  - Intergrated Clinical Oncology Network (ICON), South Brisbane, Queensland
  - Icon Cancer Care Southport, Southport, Queensland
  - Eastern Clinical Research Unit, Box Hill, Victoria
  - Eastern Health Pathology Service, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Peninsula Health, Frankston, Victoria
  - Olivia Newton John Cancer Wellness & Research Centre Austin Health, Heidelberg, Victoria
- Austria (8):
  - Ordensklinikum Linz, Barmherzige Schwestern, Linz, Upper Austria
  - Vinzenz Pathologieverbund, Linz, Upper Austria
  - Ordensklinikum Linz GmbH, Elisabethinen, Linz, Upper Austria
  - Paracelsus Medical University, SALK, Salzburg
  - Isotopix-Ambulatorium fur Nuklearmedizin, Vienna
  - Medical University of Vienna, Vienna
  - Medizinische Universitat Wien, Vienna
  - Diagnosezentrum Meidling, Vienna
- Belgium (3):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Algemeen Ziekenhuis Sint-Lucas, Ghent
  - UZ Leuven, Campus Gasthuisberg, Leuven
- Brazil (4):
  - Hospital de Caridade de Ijui, Ijuí, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre-HCPA, Porto Alegre, Rio Grande do Sul
  - Fundacao Pio XII-Hospital de Cancer de Barretos, Barretos, São Paulo
  - Fundacao Doutor Amaral Carvalho, Jaú, São Paulo
- France (8):
  - ICO-Site Paul Papin, Angers
  - CHRUBesangon-H6pital Jean Minjoz, Besançon
  - Institut Bergonie, Service d'Oncologie, Bordeaux
  - Centre Hospitalier Departemental Les Oudairies, La Roche-sur-Yon
  - Clinique Victor Hugo-Centre Jean Bernard, Le Mans
  - Institut de Cancerologie Strasbourg Europe, Strasbourg
  - Hopital Foch Service Oncologie, Suresnes
  - Institut Gustave Roussy, Villejuif
- Germany (7):
  - Universitaetsklinikum Essen, Essen
  - Medizinische Hochschule Hannover, Hanover
  - Medizinische Fakultat Mannheim der Universitat Heidelberg, Mannheim
  - Universitatsklinikum Munster, Münster
  - Studienpraxis Urologie, Nürtingen
  - Universitatsklinikum Tubingen, Tübingen
  - Universitaetsklinikum Wuerzburg, Würzburg
- Hungary (4):
  - Semmelweis Egyetem, Budapest
  - Orszagos Onkologiai Intezet, "C" Belgyogyaszati-Onkologiai es Klinikai Farmakogogiai Osztaly, Budapest
  - Debreceni Egyetem, Debrecen
  - Szabolcs- Szatmar-Bereg Megyei Korhazak es Egyetemi Oktato Korhaz, Nyíregyháza
- Italy (10):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola, Forli - Cesena
  - Azienda Ospedaliera San Camillo Forlanini, Roma, ROME
  - Azienda Ospedaliero-Universitaria S. Luigi Gonzaga-SCDU Oncologia Medica, Orbassano, Torino/piemonte
  - AULSS3 Serenissima - Ospedale dell'Angelo - Oncologia Medica, Mestre, Venezia
  - Azienda Socio Sanitaria Territoriale di Cremona (Istituti Ospitalieri di Cremona), Cremona
  - SD Oncologia Clinica Sperimentale di Uro-Ginecologia, Napoli
  - IOV - Istituto Oncologico Veneto IRCCS - U.O. Oncologia Medica 1, Padua
  - Azienda Ospedaliero Universitari di Parma - U.O. Oncologia Medica, Parma
  - Azienda Ospedaliero Universitaria di Parma - U.O. Oncologia Medica, Parma
  - Azienda Ospedaliero Universitaria Citta della Salute e della Scienza di Torino, Torino
- Radboud UMC, Nijmegen, THE Netherlands, Netherlands
- Poland (2):
  - Szpital Specjalistyczny W Brzozowie, Podkarpacki Osrodek Onkologiczny Im.Ks.B.Markiewicza, Brzozów
  - Swietokrzyskie Centrum Onkologii Samodzielny Publiczny Zaklad Opieki Zdrowotnej, Kielce
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Pusan National University Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Spain (7):
  - Hospital Virgen de la Victoria, Málaga, Malga
  - Clinica Universidad de Navarra-Oncology Service, Pamplona, Navarre
  - Hospital General Vall D'Hebron-Oncology Service, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Quironsalud Madrid-Oncology Service, Madrid
  - Instituto Valenciano de Oncologia (IVO-FINCIVO), Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia
- United Kingdom (3):
  - Mount Vernon Hospital, Northwood, Middlesex
  - The Institute of Cancer Research, The Royal Marsden NHS Foundation Trust , Sycamore House, Sutton, Surrey
  - Addenbrookes Hospital, Cambridge

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Mehra N, Fizazi K, de Bono JS, Barthelemy P, Dorff T, Stirling A, Machiels JP, Bimbatti D, Kilari D, Dumez H, Buttigliero C, van Oort IM, Castro E, Chen HC, Di Santo N, DeAnnuntis L, Healy CG, Scagliotti GV. Talazoparib, a Poly(ADP-ribose) Polymerase Inhibitor, for Metastatic Castration-resistant Prostate Cancer and DNA Damage Response Alterations: TALAPRO-1 Safety Analyses. Oncologist. 2022 Oct 1;27(10):e783-e795. doi: 10.1093/oncolo/oyac172. PMID 36124924
- [Derived] de Bono JS, Mehra N, Scagliotti GV, Castro E, Dorff T, Stirling A, Stenzl A, Fleming MT, Higano CS, Saad F, Buttigliero C, van Oort IM, Laird AD, Mata M, Chen HC, Healy CG, Czibere A, Fizazi K. Talazoparib monotherapy in metastatic castration-resistant prostate cancer with DNA repair alterations (TALAPRO-1): an open-label, phase 2 trial. Lancet Oncol. 2021 Sep;22(9):1250-1264. doi: 10.1016/S1470-2045(21)00376-4. Epub 2021 Aug 10. PMID 34388386
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=MDV3800-06

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with measurable soft tissue disease as per response evaluation criteria in solid tumors (RECIST) 1.1 and progressive metastatic castration-resistant prostate cancer (CRPC) and deoxyribonucleic acid (DNA) damage repair deficiencies, who previously received 1 to 2 taxane-based chemotherapy, and progressed on at least 1 line of novel hormonal therapy (enzalutamide and/or abiraterone acetate/prednisone) were enrolled.
Groups:
- Talazoparib: Participants received talazoparib 1 milligram per day (mg/day) orally until radiographic progression that was determined by independent central review, unacceptable toxicity, withdrawal of consent, or death. Talazoparib was continued upon disease progression only if, in the opinion of the investigator the participant was clinically benefitting, no new concurrent systemic therapy was initiated, and the sponsor was notified. Maximum duration of treatment was approximately 36 months.
Period: Overall Study
Arm/Group | Talazoparib
Started | 128
Completed | 127
Not Completed | 1
Not completed — Progressive Disease | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of talazoparib including participants enrolled prior to protocol amendment 3 with non-measurable disease and with deoxyribonucleic acid damage response (DDR) deficiencies which was likely or might sensitized the tumor to poly adenosine diphosphate-ribose polymerase (PARP) inhibition as assessed using an expanded DDR gene panel.
Arm/Group | Talazoparib
Number analyzed (Participants) | 127
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Mean | 68.16 (8.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 127
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 106
  Unknown or Not Reported | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 110
  More than one race | 0
  Unknown or Not Reported | 10

OUTCOME MEASURES:

1. Primary Outcome: Best Objective Response Rate (ORR)
Description: Best ORR was defined as the percentage of participants with best overall soft tissue response of complete response (CR) or partial response (PR) as per RECIST1.1 by an independent central review. RECIST 1.1 criteria, CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than 10 millimeter (mm). Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (less than 10 mm short axis); PR: at least 30 percent (%) decrease in sum of diameters of target lesions taking as reference baseline sum diameters.
Time Frame: From first dose of study drug to best overall soft tissue response CR or PR (maximum duration of 25 months)
Population: DDR deficient measurable disease population included all enrolled participants who had measurable soft tissue disease at screening by investigator assessment, had DDR deficiencies likely to sensitize to PARP inhibitor therapy, and received at least 1 dose of talazoparib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Talazoparib
Number analyzed (Participants) | 104
Percentage of participants | 29.8 [21.2 to 39.6]

2. Secondary Outcome: Time to Objective Response
Description: Time to objective response was defined as the time from first dose of talazoparib to the first objective evidence of soft tissue response with no evidence of confirmed bone disease progression on bone scan per prostate cancer working Group 3 (PCWG3). Soft tissue response is defined as a best overall response of CR or PR per RECIST 1.1 by independent central review. RECIST 1.1 criteria, CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than 10 mm. Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (less than 10 mm short axis); PR: at least 30 % decrease in sum of diameters of target lesions taking as reference baseline sum diameters.
Time Frame: From first dose of study drug to first objective response (maximum duration of 25 months)
Population: DDR deficient measurable disease population included all enrolled participants who had measurable soft tissue disease at screening by investigator assessment, had DDR deficiencies likely to sensitize to PARP inhibitor therapy, and received at least 1 dose of talazoparib and participants who achieved a confirmed CR or PR without documentation of confirmed bone progression.
Measure: Median (Full Range); unit: Months
Arm/Group | Talazoparib
Number analyzed (Participants) | 31
Months | 3.4 [1.6 to 7.5]

3. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the first objective evidence of soft tissue response (CR or PR, whichever is earlier) per RECIST 1.1 and no evidence of confirmed bone disease progression per PCWG3 to the date of first objective evidence of radiographic progression or death due to any cause without evidence of radiographic progression, whichever occurs first. RECIST 1.1 criteria, CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than 10 mm. Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (less than 10 mm short axis); PR: at least 30 % decrease in sum of diameters of target lesions taking as reference baseline sum diameters.
Time Frame: From the first objective evidence of soft tissue response (CR or PR, whichever is earlier) to radiographic progression or death due to any cause without evidence of radiographic progression, whichever occurs first (maximum duration of 25 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Talazoparib
Number analyzed (Participants) | 31
Months | 12.8 [6.5 to NA] — Upper limit of 95% confidence interval (CI) was not estimable as there were less number of participants with an event.

4. Secondary Outcome: Percentage of Participants With Prostate-Specific Antigen (PSA) Response of Greater Than or Equal to (>=) 50 Percentage (%)
Description: Percentage of participants with PSA response of >= 50% was reported in this outcome measure. PSA response was calculated as a decline from baseline PSA (ng/mL) by at least 50% measured by central laboratory.
Time Frame: From the date of first dose of study treatment until confirmed PSA progression or start of new anticancer treatment given after the first dose of study treatment (maximum duration of 25 months)
Population: DDR deficient measurable disease population included all enrolled participants who had measurable soft tissue disease at screening by investigator assessment, had DDR deficiencies likely to sensitize to PARP inhibitor therapy, and received at least 1 dose of talazoparib. Here ''Number of participants analyzed'' signifies number of participants evaluable data for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Talazoparib
Number analyzed (Participants) | 96
Percentage of participants | 45.8 [35.6 to 56.3]

5. Secondary Outcome: Percentage of Participants With Conversion of Circulating Tumor Cell (CTC) Count
Description: Percentage of participants with conversion of CTC count was defined as percentage of participants with a CTC count >= 5 CTC per 7.5 milliliter (mL) of blood at baseline that decreased to < 5 CTC per 7.5 mL of blood any time on study.
Time Frame: Baseline to anytime on study during final analysis of the outcome measure, up to maximum duration of 25 months
Population: All participants with a baseline CTC assessment and at least 1 post-baseline CTC assessment from the DDR deficient measurable disease population. Participants with a CTC count <5 per 7.5 mL of blood at baseline were not analyzed for this conversion outcome measure. Here, "Number of participants analyzed'' signifies number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Talazoparib
Number analyzed (Participants) | 33
Percentage of participants | 63.6 [45.1 to 79.6]

6. Secondary Outcome: Percentage of Participants With a Null CTC Count
Description: Percentage of participants with a null CTC count was defined as percentage of participants with CTC count >=1 CTC per 7.5 mL of blood at baseline that decreased to CTC = 0 per 7.5 mL of blood any time on study.
Time Frame: Baseline to anytime on study during final analysis of the outcome measure, up to maximum duration of 25 months
Population: All participants with a baseline CTC assessment and at least 1 post-baseline CTC assessment from the DDR deficient measurable disease population. Participants with a CTC count 0 per 7.5 mL of blood at baseline were not analyzed for this outcome measure.Here, "Number of participants analyzed'' signifies number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Talazoparib
Number analyzed (Participants) | 45
Percentage of participants | 53.3 [37.9 to 68.3]

7. Secondary Outcome: Percentage of Participants With Baseline CTC Count <5 CTC Showed Increased CTC Counts at Any Time on Study
Description: Percentage of participants with CTC count <5 CTC per 7.5 mL of blood at baseline those who showed an increased CTC count, compared to baseline, any time on study was reported in this study.
Time Frame: Baseline to anytime on study during final analysis of the outcome measure, up to maximum duration of 25 months
Population: All participants with a baseline CTC assessment and at least 1 post-baseline CTC assessment from the DDR deficient measurable disease population. Here, "Number of participants analyzed'' signifies number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Talazoparib
Number analyzed (Participants) | 29
Percentage of participants | 37.9 [20.7 to 57.7]

8. Secondary Outcome: Time to Prostate-Specific Antigen (PSA) Progression
Description: Time to PSA progression was defined as the time from first dose of study treatment to the date of PSA progression, which was subsequently confirmed. The time from first dose of talazoparib to the date that a >=25% increase in PSA with an absolute increase of >=2micogram per liter (2 nanogram per mL) above the nadir (or baseline for participants with no PSA decline) was documented, confirmed by a second consecutive PSA value obtained >=3 weeks (21 days) later. Kaplan-Meier method was used for analysis.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Talazoparib
Number analyzed (Participants) | 104
Months | 9.2 [5.6 to 11.1]

9. Secondary Outcome: Radiographic Progression-Free Survival (PFS)
Description: Radiographic PFS was defined as the time from date of first dose of talazoparib to first objective evidence of radiographic progression as assessed in soft tissue per modified RECIST 1.1 or confirmed progression in bone per PCWG3 guidelines by independent central review or death without documented radiographic progression, whichever occurs first.
Time Frame: From date of first dose of study drug to first objective evidence of radiographic progression or death without documented radiographic progression, whichever occurs first (maximum duration of 25 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Talazoparib
Number analyzed (Participants) | 104
Months | 5.6 [3.7 to 8.8]

10. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from start date (the date of first dose of treatment) to the date of death due to any cause. Participants who had not died were censored at the date of last contact. Kaplan-Meier method was used for analysis.
Time Frame: From first dose of study treatment up to death due to any cause during study or date of last contact (approximately 36 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Talazoparib
Number analyzed (Participants) | 104
Months | 16.9 [13.0 to 20.7]

11. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AEs included both serious AEs and all non-serious AEs. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: First dose of study drug up to 28 days after last dose of study drug (study treatment was approximately for 36 months, safety follow up to approximately 37 months)
Population: Safety population included all participants who received at least 1 dose of talazoparib including participants enrolled prior to amendment 3 with non-measurable disease and/or with DDR deficiencies, which may sensitize the tumor to PARP inhibition as assessed using an expanded DDR gene panel.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib
Number analyzed (Participants) | 127
Participants | 125

12. Secondary Outcome: Number of Participants With Permanent Treatment Discontinuation Due to Adverse Events
Description: Treatment discontinuation was defined as permanent cessation of study drug treatment administration.
Time Frame: During study treatment (approximately up to 36 months)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib
Number analyzed (Participants) | 127
Participants | 21

13. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: Vital sign abnormalities criteria included: 1) Systolic blood pressure (SBP) in millimeters of mercury (mmHg): absolute result greater than (>) 180 mmHg and increase from baseline greater than or equal to (>=) 40 mmHg or absolute result < 90 mmHg and decrease from baseline > 30 mmHg; 2) Diastolic blood pressure (DBP) (mmHg): absolute result > 110 mmHg and increase from baseline >= 30 mmHg or absolute result < 50 mmHg and decrease from baseline > 20 mmHg or >= 20 mmHg increase from baseline; 3) Heart rate in beats per minutes (bpm): absolute result < 50 bpm and decrease from baseline > 20 bpm or absolute result > 120 bpm and increase from baseline > 30 bpm; Weight in kilogram: > 10% decrease from baseline.
Time Frame: During study treatment (approximately up to 36 months)
Population: Safety population included all participants who received at least 1 dose of talazoparib including participants enrolled prior to amendment 3 with non-measurable disease and/or with DDR deficiencies, which may sensitize the tumor to PARP inhibition as assessed using an expanded DDR gene panel. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies those participants who were evaluable at specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib
Number analyzed (Participants) | 125
Participants
  SBP: Absolute result > 180 mm Hg and increase from baseline >= 40 mm Hg | 0
  SBP: Absolute result < 90 mm Hg and decrease from baseline > 30 mm Hg | 0
  DBP: Absolute result > 110 mm Hg and increase from baseline >= 30 mm Hg | 0
  DBP: Absolute result < 50 mm Hg and decrease from baseline > 20 mm Hg | 0
  DBP: >= 20 mm Hg increase from baseline | 17
  Heart rate: Absolute result < 50 bpm and decrease from baseline > 20 bpm | 0
  Heart rate: Absolute result > 120 bpm and increase from baseline > 30 bpm | 2
  Weight: > 10% decrease from baseline: number analyzed (Participants) | 124
  Weight: > 10% decrease from baseline | 0

14. Secondary Outcome: Number of Participants With Shift in Laboratory Parameter Values (Hematology) From Grade Less Than Equal to (<=) 2 at Baseline to Grade 3 or 4 Post-baseline
Description: Hematology parameters included anemia, hemoglobin increased, lymphocyte count decreased, lymphocyte count increased, neutrophil count decreased, platelet count decreased, Leukocytosis and white blood cell decreased. Severity was graded as Grade 1: asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated; Grade 2: moderate, minimal, local or non-invasive intervention indicated, limiting age-appropriate instrumental activities of daily life (ADL); Grade 3: severe or medically significant but not immediately life-threatening, hospitalization or prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4: life-threatening consequence, urgent intervention indicated; Grade 5: death related to AE.
Time Frame: During study treatment (approximately up to 36 months)
Population: Safety population included all participants who received at least 1 dose of talazoparib including participants enrolled prior to amendment 3 with non-measurable disease and/or with DDR deficiencies, which may sensitize the tumor to PARP inhibition as assessed using an expanded DDR gene panel. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib
Number analyzed (Participants) | 125
Participants
  Anemia | 30
  Hemoglobin increased | 1
  Lymphocyte count decreased | 23
  Lymphocyte count increased | 0
  Neutrophil count decreased | 11
  Platelet count decreased | 3
  White blood cell decreased | 5
  Leukocytosis | 0

15. Secondary Outcome: Number of Participants With Shift in Laboratory Parameter Values (Chemistry) From Grade <=2 at Baseline to Grade 3 or 4 Post-baseline
Description: Chemistry parameters:alanine aminotransferase increased(inc), alkaline phosphatase inc, aspartate aminotransferase inc, blood bilirubin inc, chronic kidney disease, creatinine inc, gamma-glutamyl transferase (GGT) inc, hypercalcemia, Hyperglycemia, hyperkalemia, hypermagnesemia, hypocalcemia, Hyponatremia, hypoglycemia, hypokalemia, hypomagnesemia, hypernatremia, Hypoalbuminemia and hypophosphatemia. Severity was graded as Grade(G)1: asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated; G2:moderate, minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental ADL; G3:severe or medically significant but not immediately life-threatening, hospitalization or prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; G4:life-threatening consequence, urgent intervention indicated; G5: death related to AEs.
Time Frame: During study treatment (approximately up to 36 months)
Population: Safety population included all participants who received at least 1 dose of talazoparib including participants enrolled prior to amendment 3 with non-measurable disease and/or with DDR deficiencies, which may sensitize the tumor to PARP inhibition as assessed using an expanded DDR gene panel. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants evaluable at specific rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib
Number analyzed (Participants) | 126
Participants
  Alanine aminotransferase increased | 0
  Alkaline phosphatase increased | 9
  Aspartate aminotransferase increased | 0
  Blood bilirubin increased | 0
  Chronic kidney disease | 2
  Creatinine increased | 1
  GGT increased: number analyzed (Participants) | 53
  GGT increased | 3
  Hypercalcemia | 0
  Hyperglycemia | 5
  Hyperkalemia | 4
  Hypermagnesemia | 1
  Hypernatremia | 0
  Hypoalbuminemia | 0
  Hypocalcemia | 4
  Hypoglycemia | 0
  Hypokalemia | 0
  Hypomagnesemia | 1
  Hyponatremia | 3
  Hypophosphatemia | 2

16. Secondary Outcome: Number of Participants With Dose Modification
Description: Number of participants with dose modification due to adverse events was reported.
Time Frame: During study treatment (approximately up to 36 months)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib
Number analyzed (Participants) | 127
Participants | 37

17. Secondary Outcome: Time to Deterioration in Pain Symptom Scores
Description: Time deterioration is based on BPI-SF question 3: "Please rate your pain by marking the box beside the number that best describes your pain at its worst in the last 24 hours." Pain intensity was to be answered on a range of 0 to 10, where 0 corresponded to no pain and 10 worst pain. Time to this event is defined as the time from the date of first dose of study treatment to onset of pain progression, where pain progression is defined as a 2-point or more increase from baseline in the question 3 score. Kaplan-Meier method was used for analysis. Average of all assessments visits is reported in this outcome measure.
Time Frame: Baseline till final analysis of the outcome measure, up to maximum duration of 25 months
Population: All participants from the DDR deficient measurable disease population with a baseline PRO assessment and at least 1 post-baseline PRO assessment prior to the end of treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Talazoparib
Number analyzed (Participants) | 97
Months | NA [NA to NA] — Median and 95 % confidence interval could not be estimated due to insufficient number of participants with event.

18. Secondary Outcome: Change From Baseline in Participant Reported Pain Scores Per BPI-SF Question 3
Description: BPI-SF is an 11-item self-report questionnaire that is designed to assess the severity and impact of pain on daily functions. BPI-SF have 4 questions that assess pain intensity (worst, least, average, right now) and 7 questions that assess impact of pain on daily functions (general activity, mood, walking ability, normal work, relations with other people, sleep, enjoyment of life). Each question is answered on a scale ranging from 0 to 10; '0=No pain and 10=Pain as bad as you can imagine'. Measure can be scored by item, with lower scores being indicative of less pain or pain interference. BPI-SF question 3 was related to participant experiencing pain at its worst in last 24 hours, score range 0 to 10, where large values corresponded to worse outcomes.
Time Frame: Baseline, Week 1, 3, 5, 7, 9, 13, 17, 21, 25, 37, 49, 61, 73, 85, Follow-up Visit (28 days after last dose) [maximum duration of 25 months]
Population: All participants from the DDR deficient measurable disease population with a baseline PRO assessment and at least 1 post-baseline PRO assessment prior to the end of treatment. All participants reported under 'Overall Number of Participants Analyzed' contributed data to the table; however, may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants evaluable for specified time points.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Talazoparib
Number analyzed (Participants) | 97
Units on a scale
  Change at Week 1: number analyzed (Participants) | 0
  Change at Week 3: number analyzed (Participants) | 70
  Change at Week 3 | -0.51 (2.04)
  Change at Week 5: number analyzed (Participants) | 72
  Change at Week 5 | -1.39 (2.55)
  Change at Week 7: number analyzed (Participants) | 61
  Change at Week 7 | -1.20 (2.89)
  Change at Week 9: number analyzed (Participants) | 63
  Change at Week 9 | -1.25 (2.38)
  Change at Week 13: number analyzed (Participants) | 55
  Change at Week 13 | -0.85 (2.51)
  Change at Week 17: number analyzed (Participants) | 54
  Change at Week 17 | -1.06 (2.73)
  Change at Week 21: number analyzed (Participants) | 44
  Change at Week 21 | -0.89 (2.77)
  Change at Week 25: number analyzed (Participants) | 44
  Change at Week 25 | -1.14 (3.14)
  Change at Week 37: number analyzed (Participants) | 27
  Change at Week 37 | -1.00 (2.30)
  Change at Week 49: number analyzed (Participants) | 17
  Change at Week 49 | -1.53 (3.50)
  Change at Week 61: number analyzed (Participants) | 12
  Change at Week 61 | -2.50 (3.42)
  Change at Week 73: number analyzed (Participants) | 5
  Change at Week 73 | -2.80 (5.17)
  Change at Week 85: number analyzed (Participants) | 2
  Change at Week 85 | -5.50 (3.54)
  Change at Follow-up: number analyzed (Participants) | 24
  Change at Follow-up | -0.25 (3.21)

19. Secondary Outcome: Change From Baseline in European Quality of Life 5-Domain 5-Level Scale (EQ-5D-5L) Visual Analogue Scores (VAS)
Description: The EQ-5D VAS score was a participant rated questionnaire where participants rated how they felt at assessment visit on a vertical VAS that ranged from 0 (worst imaginable health state) to 100 (best imaginable health state), with higher scores indicating a better health condition.
Time Frame: Baseline, Week 1, 3, 5,7, 9, 13, 17, 21, 25, 37, 49, 61, 73, 85, 97, Follow-up Visit (28 days after last dose) [maximum duration of 25 months]
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Talazoparib
Number analyzed (Participants) | 97
Units on a scale
  Change at Week 1: number analyzed (Participants) | 0
  Change at Week 3: number analyzed (Participants) | 89
  Change at Week 3 | 4.16 (17.25)
  Change at Week 5: number analyzed (Participants) | 93
  Change at Week 5 | 4.44 (17.26)
  Change at Week 7: number analyzed (Participants) | 84
  Change at Week 7 | 6.61 (17.20)
  Change at Week 9: number analyzed (Participants) | 88
  Change at Week 9 | 6.18 (20.21)
  Change at Week 13: number analyzed (Participants) | 71
  Change at Week 13 | 7.68 (16.85)
  Change at Week 17: number analyzed (Participants) | 73
  Change at Week 17 | 7.84 (19.40)
  Change at Week 21: number analyzed (Participants) | 62
  Change at Week 21 | 6.63 (19.26)
  Change at Week 25: number analyzed (Participants) | 59
  Change at Week 25 | 5.34 (21.50)
  Change at Week 37: number analyzed (Participants) | 37
  Change at Week 37 | 4.65 (19.01)
  Change at Week 49: number analyzed (Participants) | 23
  Change at Week 49 | 8.96 (17.55)
  Change at Week 61: number analyzed (Participants) | 16
  Change at Week 61 | 12.75 (19.02)
  Change at Week 73: number analyzed (Participants) | 8
  Change at Week 73 | 1.25 (24.89)
  Change at Week 85: number analyzed (Participants) | 4
  Change at Week 85 | 11.50 (25.01)
  Change at Week 97: number analyzed (Participants) | 1
  Change at Week 97 | 17.00
  Change at Follow-up: number analyzed (Participants) | 30
  Change at Follow-up | -2.87 (21.55)

20. Secondary Outcome: Number of Participants With 5 Response Levels for EQ-5D-5L Mobility Domain
Description: EQ-5D-5L: participant rated assessed level of current health using 5 domains: mobility, self-care, usual activities, pain and discomfort, anxiety, and depression. EQ-5D mobility domain had 5 responses: no problem, slight problem, moderate problem, severe problem and extreme problem.
Time Frame: as for outcome 19
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib
Number analyzed (Participants) | 97
Participants
  Week 1: number analyzed (Participants) | 96
  Week 1: No Problem | 30
  Week 1: Slight Problem | 29
  Week 1: Moderate Problem | 25
  Week 1: Severe Problem | 12
  Week 1: Extreme Problem | 0
  Week 3: number analyzed (Participants) | 90
  Week 3: No Problem | 36
  Week 3: Slight Problem | 23
  Week 3: Moderate Problem | 20
  Week 3: Severe Problem | 10
  Week 3: Extreme Problem | 1
  Week 5: number analyzed (Participants) | 95
  Week 5: No Problem | 36
  Week 5: Slight Problem | 29
  Week 5: Moderate Problem | 23
  Week 5: Severe Problem | 6
  Week 5: Extreme Problem | 1
  Week 7: number analyzed (Participants) | 86
  Week 7: No Problem | 37
  Week 7: Slight Problem | 24
  Week 7: Moderate Problem | 22
  Week 7: Severe Problem | 3
  Week 7: Extreme Problem | 0
  Week 9: number analyzed (Participants) | 90
  Week 9: No Problem | 38
  Week 9: Slight Problem | 26
  Week 9: Moderate Problem | 20
  Week 9: Severe Problem | 4
  Week 9: Extreme Problem | 2
  Week 13: number analyzed (Participants) | 73
  Week 13: No Problem | 28
  Week 13: Slight Problem | 26
  Week 13: Moderate Problem | 12
  Week 13: Severe Problem | 5
  Week 13: Extreme Problem | 2
  Week 17: number analyzed (Participants) | 74
  Week 17: No Problem | 30
  Week 17: Slight Problem | 28
  Week 17: Moderate Problem | 14
  Week 17: Severe Problem | 1
  Week 17: Extreme Problem | 1
  Week 21: number analyzed (Participants) | 63
  Week 21: No Problem | 30
  Week 21: Slight Problem | 15
  Week 21: Moderate Problem | 15
  Week 21: Severe Problem | 3
  Week 21: Extreme Problem | 0
  Week 25: number analyzed (Participants) | 59
  Week 25: No Problem | 29
  Week 25: Slight Problem | 14
  Week 25: Moderate Problem | 13
  Week 25: Severe Problem | 3
  Week 25: Extreme Problem | 0
  Week 37: number analyzed (Participants) | 37
  Week 37: No Problem | 16
  Week 37: Slight Problem | 14
  Week 37: Moderate Problem | 4
  Week 37: Severe Problem | 3
  Week 37: Extreme Problem | 0
  Week 49: number analyzed (Participants) | 23
  Week 49: No Problem | 10
  Week 49: Slight Problem | 7
  Week 49: Moderate Problem | 5
  Week 49: Severe Problem | 1
  Week 49: Extreme Problem | 0
  Week 61: number analyzed (Participants) | 16
  Week 61: No Problem | 7
  Week 61: Slight Problem | 5
  Week 61: Moderate Problem | 3
  Week 61: Severe Problem | 1
  Week 61: Extreme Problem | 0
  Week 73: number analyzed (Participants) | 8
  Week 73: No Problem | 4
  Week 73: Slight Problem | 2
  Week 73: Moderate Problem | 2
  Week 73: Severe Problem | 0
  Week 73: Extreme Problem | 0
  Week 85: number analyzed (Participants) | 4
  Week 85: No Problem | 2
  Week 85: Slight Problem | 2
  Week 85: Moderate Problem | 0
  Week 85: Severe Problem | 0
  Week 85: Extreme Problem | 0
  Week 97: number analyzed (Participants) | 1
  Week 97: No Problem | 1
  Week 97: Slight Problem | 0
  Week 97: Moderate Problem | 0
  Week 97: Severe Problem | 0
  Week 97: Extreme Problem | 0
  Follow-up: number analyzed (Participants) | 30
  Follow-up: No Problem | 11
  Follow-up: Slight Problem | 8
  Follow-up: Moderate Problem | 6
  Follow-up: Severe Problem | 5
  Follow-up: Extreme Problem | 0

21. Secondary Outcome: Number of Participants With 5 Response Levels for EQ-5D-5L Self-Care Domain
Description: EQ-5D-5L: participant rated assessed level of current health using 5 domains: mobility, self-care, usual activities, pain and discomfort, anxiety, and depression. EQ-5D self-care domain had 5 responses: no problem, slight problem, moderate problem, severe problem and extreme problem.
Time Frame: as for outcome 19
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib
Number analyzed (Participants) | 97
Participants
  Week 1: number analyzed (Participants) | 95
  Week 1: No Problem | 65
  Week 1: Slight Problem | 18
  Week 1: Moderate Problem | 9
  Week 1: Severe Problem | 3
  Week 1: Extreme Problem | 0
  Week 3: number analyzed (Participants) | 90
  Week 3: No Problem | 63
  Week 3: Slight Problem | 17
  Week 3: Moderate Problem | 8
  Week 3: Severe Problem | 2
  Week 3: Extreme Problem | 0
  Week 5: number analyzed (Participants) | 95
  Week 5: No Problem | 62
  Week 5: Slight Problem | 20
  Week 5: Moderate Problem | 12
  Week 5: Severe Problem | 1
  Week 5: Extreme Problem | 0
  Week 7: number analyzed (Participants) | 85
  Week 7: No Problem | 59
  Week 7: Slight Problem | 14
  Week 7: Moderate Problem | 12
  Week 7: Severe Problem | 0
  Week 7: Extreme Problem | 0
  Week 9: number analyzed (Participants) | 90
  Week 9: No Problem | 64
  Week 9: Slight Problem | 15
  Week 9: Moderate Problem | 8
  Week 9: Severe Problem | 2
  Week 9: Extreme Problem | 1
  Week 13: number analyzed (Participants) | 73
  Week 13: No Problem | 51
  Week 13: Slight Problem | 14
  Week 13: Moderate Problem | 3
  Week 13: Severe Problem | 4
  Week 13: Extreme Problem | 1
  Week 17: number analyzed (Participants) | 74
  Week 17: No Problem | 55
  Week 17: Slight Problem | 13
  Week 17: Moderate Problem | 4
  Week 17: Severe Problem | 2
  Week 17: Extreme Problem | 0
  Week 21: number analyzed (Participants) | 63
  Week 21: No Problem | 44
  Week 21: Slight Problem | 12
  Week 21: Moderate Problem | 5
  Week 21: Severe Problem | 2
  Week 21: Extreme Problem | 0
  Week 25: number analyzed (Participants) | 59
  Week 25: No Problem | 39
  Week 25: Slight Problem | 13
  Week 25: Moderate Problem | 7
  Week 25: Severe Problem | 0
  Week 25: Extreme Problem | 0
  Week 37: number analyzed (Participants) | 37
  Week 37: No Problem | 25
  Week 37: Slight Problem | 10
  Week 37: Moderate Problem | 2
  Week 37: Severe Problem | 0
  Week 37: Extreme Problem | 0
  Week 49: number analyzed (Participants) | 23
  Week 49: No Problem | 18
  Week 49: Slight Problem | 4
  Week 49: Moderate Problem | 1
  Week 49: Severe Problem | 0
  Week 49: Extreme Problem | 0
  Week 61: number analyzed (Participants) | 16
  Week 61: No Problem | 11
  Week 61: Slight Problem | 5
  Week 61: Moderate Problem | 0
  Week 61: Severe Problem | 0
  Week 61: Extreme Problem | 0
  Week 73: number analyzed (Participants) | 8
  Week 73: No Problem | 7
  Week 73: Slight Problem | 1
  Week 73: Moderate Problem | 0
  Week 73: Severe Problem | 0
  Week 73: Extreme Problem | 0
  Week 85: number analyzed (Participants) | 4
  Week 85: No Problem | 4
  Week 85: Slight Problem | 0
  Week 85: Moderate Problem | 0
  Week 85: Severe Problem | 0
  Week 85: Extreme Problem | 0
  Week 97: number analyzed (Participants) | 1
  Week 97: No Problem | 1
  Week 97: Slight Problem | 0
  Week 97: Moderate Problem | 0
  Week 97: Severe Problem | 0
  Week 97: Extreme Problem | 0
  Follow-up: number analyzed (Participants) | 30
  Follow-up: No Problem | 19
  Follow-up: Slight Problem | 3
  Follow-up: Moderate Problem | 7
  Follow-up: Severe Problem | 1
  Follow-up: Extreme Problem | 0

22. Secondary Outcome: Number of Participants With 5 Response Levels for EQ-5D-5L Usual Activity Domain
Description: EQ-5D-5L: participant rated assessed level of current health using 5 domains: mobility, self-care, usual activities, pain and discomfort, anxiety, and depression. EQ-5D usual activities domain had 5 responses: no problem, slight problem, moderate problem, severe problem and extreme problem.
Time Frame: as for outcome 19
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib
Number analyzed (Participants) | 97
Participants
  Week 1: number analyzed (Participants) | 96
  Week 1: No Problem | 33
  Week 1: Slight Problem | 30
  Week 1: Moderate Problem | 19
  Week 1: Severe Problem | 10
  Week 1: Extreme Problem | 4
  Week 3: number analyzed (Participants) | 90
  Week 3: No Problem | 33
  Week 3: Slight Problem | 26
  Week 3: Moderate Problem | 22
  Week 3: Severe Problem | 8
  Week 3: Extreme Problem | 1
  Week 5: number analyzed (Participants) | 95
  Week 5: No Problem | 36
  Week 5: Slight Problem | 30
  Week 5: Moderate Problem | 21
  Week 5: Severe Problem | 4
  Week 5: Extreme Problem | 4
  Week 7: number analyzed (Participants) | 85
  Week 7: No Problem | 34
  Week 7: Slight Problem | 24
  Week 7: Moderate Problem | 22
  Week 7: Severe Problem | 3
  Week 7: Extreme Problem | 2
  Week 9: number analyzed (Participants) | 90
  Week 9: No Problem | 41
  Week 9: Slight Problem | 26
  Week 9: Moderate Problem | 15
  Week 9: Severe Problem | 5
  Week 9: Extreme Problem | 3
  Week 13: number analyzed (Participants) | 73
  Week 13: No Problem | 36
  Week 13: Slight Problem | 22
  Week 13: Moderate Problem | 10
  Week 13: Severe Problem | 2
  Week 13: Extreme Problem | 3
  Week 17: number analyzed (Participants) | 74
  Week 17: No Problem | 36
  Week 17: Slight Problem | 21
  Week 17: Moderate Problem | 14
  Week 17: Severe Problem | 2
  Week 17: Extreme Problem | 1
  Week 21: number analyzed (Participants) | 63
  Week 21: No Problem | 35
  Week 21: Slight Problem | 13
  Week 21: Moderate Problem | 12
  Week 21: Severe Problem | 2
  Week 21: Extreme Problem | 1
  Week 25: number analyzed (Participants) | 59
  Week 25: No Problem | 29
  Week 25: Slight Problem | 12
  Week 25: Moderate Problem | 12
  Week 25: Severe Problem | 6
  Week 25: Extreme Problem | 0
  Week 37: number analyzed (Participants) | 37
  Week 37: No Problem | 17
  Week 37: Slight Problem | 10
  Week 37: Moderate Problem | 7
  Week 37: Severe Problem | 3
  Week 37: Extreme Problem | 0
  Week 49: number analyzed (Participants) | 23
  Week 49: No Problem | 11
  Week 49: Slight Problem | 5
  Week 49: Moderate Problem | 6
  Week 49: Severe Problem | 1
  Week 49: Extreme Problem | 0
  Week 61: number analyzed (Participants) | 16
  Week 61: No Problem | 8
  Week 61: Slight Problem | 4
  Week 61: Moderate Problem | 3
  Week 61: Severe Problem | 1
  Week 61: Extreme Problem | 0
  Week 73: number analyzed (Participants) | 8
  Week 73: No Problem | 6
  Week 73: Slight Problem | 0
  Week 73: Moderate Problem | 2
  Week 73: Severe Problem | 0
  Week 73: Extreme Problem | 0
  Week 85: number analyzed (Participants) | 4
  Week 85: No Problem | 2
  Week 85: Slight Problem | 2
  Week 85: Moderate Problem | 0
  Week 85: Severe Problem | 0
  Week 85: Extreme Problem | 0
  Week 97: number analyzed (Participants) | 1
  Week 97: No Problem | 1
  Week 97: Slight Problem | 0
  Week 97: Moderate Problem | 0
  Week 97: Severe Problem | 0
  Week 97: Extreme Problem | 0
  Follow-up: number analyzed (Participants) | 30
  Follow-up: No Problem | 10
  Follow-up: Slight Problem | 10
  Follow-up: Moderate Problem | 5
  Follow-up: Severe Problem | 5
  Follow-up: Extreme Problem | 0

23. Secondary Outcome: Number of Participants With 5 Response Levels for EQ-5D-5L Pain and Discomfort Domain
Description: EQ-5D-5L: participant rated assessed level of current health using 5 domains: mobility, self-care, usual activities, pain and discomfort, anxiety, and depression. EQ-5D pain and discomfort domain had 5 responses: no problem, slight problem, moderate problem, severe problem and extreme problem.
Time Frame: as for outcome 19
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib
Number analyzed (Participants) | 97
Participants
  Week 1: number analyzed (Participants) | 96
  Week 1: No Problem | 15
  Week 1: Slight Problem | 35
  Week 1: Moderate Problem | 30
  Week 1: Severe Problem | 16
  Week 1: Extreme Problem | 0
  Week 3: number analyzed (Participants) | 90
  Week 3: No Problem | 25
  Week 3: Slight Problem | 25
  Week 3: Moderate Problem | 32
  Week 3: Severe Problem | 8
  Week 3: Extreme Problem | 0
  Week 5: number analyzed (Participants) | 95
  Week 5: No Problem | 30
  Week 5: Slight Problem | 27
  Week 5: Moderate Problem | 29
  Week 5: Severe Problem | 9
  Week 5: Extreme Problem | 0
  Week 7: number analyzed (Participants) | 85
  Week 7: No Problem | 26
  Week 7: Slight Problem | 32
  Week 7: Moderate Problem | 23
  Week 7: Severe Problem | 4
  Week 7: Extreme Problem | 0
  Week 9: number analyzed (Participants) | 90
  Week 9: No Problem | 34
  Week 9: Slight Problem | 29
  Week 9: Moderate Problem | 21
  Week 9: Severe Problem | 6
  Week 9: Extreme Problem | 0
  Week 13: number analyzed (Participants) | 73
  Week 13: No Problem | 23
  Week 13: Slight Problem | 33
  Week 13: Moderate Problem | 12
  Week 13: Severe Problem | 3
  Week 13: Extreme Problem | 2
  Week 17: number analyzed (Participants) | 74
  Week 17: No Problem | 27
  Week 17: Slight Problem | 25
  Week 17: Moderate Problem | 17
  Week 17: Severe Problem | 5
  Week 17: Extreme Problem | 0
  Week 21: number analyzed (Participants) | 63
  Week 21: No Problem | 24
  Week 21: Slight Problem | 19
  Week 21: Moderate Problem | 17
  Week 21: Severe Problem | 2
  Week 21: Extreme Problem | 1
  Week 25: number analyzed (Participants) | 59
  Week 25: No Problem | 22
  Week 25: Slight Problem | 17
  Week 25: Moderate Problem | 17
  Week 25: Severe Problem | 3
  Week 25: Extreme Problem | 0
  Week 37: number analyzed (Participants) | 37
  Week 37: No Problem | 12
  Week 37: Slight Problem | 12
  Week 37: Moderate Problem | 10
  Week 37: Severe Problem | 3
  Week 37: Extreme Problem | 0
  Week 49: number analyzed (Participants) | 23
  Week 49: No Problem | 11
  Week 49: Slight Problem | 3
  Week 49: Moderate Problem | 7
  Week 49: Severe Problem | 2
  Week 49: Extreme Problem | 0
  Week 61: number analyzed (Participants) | 16
  Week 61: No Problem | 6
  Week 61: Slight Problem | 5
  Week 61: Moderate Problem | 5
  Week 61: Severe Problem | 0
  Week 61: Extreme Problem | 0
  Week 73: number analyzed (Participants) | 8
  Week 73: No Problem | 2
  Week 73: Slight Problem | 4
  Week 73: Moderate Problem | 1
  Week 73: Severe Problem | 1
  Week 73: Extreme Problem | 0
  Week 85: number analyzed (Participants) | 4
  Week 85: No Problem | 2
  Week 85: Slight Problem | 2
  Week 85: Moderate Problem | 0
  Week 85: Severe Problem | 0
  Week 85: Extreme Problem | 0
  Week 97: number analyzed (Participants) | 1
  Week 97: No Problem | 0
  Week 97: Slight Problem | 1
  Week 97: Moderate Problem | 0
  Week 97: Severe Problem | 0
  Week 97: Extreme Problem | 0
  Follow-up: number analyzed (Participants) | 30
  Follow-up: No Problem | 9
  Follow-up: Slight Problem | 8
  Follow-up: Moderate Problem | 9
  Follow-up: Severe Problem | 4
  Follow-up: Extreme Problem | 0

24. Secondary Outcome: Number of Participants With 5 Response Levels for EQ-5D-5L Anxiety and Depression Domain
Description: EQ-5D-5L: participant rated assessed level of current health using 5 domains: mobility, self-care, usual activities, pain and discomfort, anxiety, and depression. EQ-5D anxiety and depression domain had 5 responses: no problem, slight problem, moderate problem, severe problem and extreme problem.
Time Frame: as for outcome 19
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib
Number analyzed (Participants) | 97
Participants
  Week 1: number analyzed (Participants) | 96
  Week 1: No Problem | 48
  Week 1: Slight Problem | 30
  Week 1: Moderate Problem | 18
  Week 1: Severe Problem | 0
  Week 1: Extreme Problem | 0
  Week 3: number analyzed (Participants) | 90
  Week 3: No Problem | 45
  Week 3: Slight Problem | 27
  Week 3: Moderate Problem | 17
  Week 3: Severe Problem | 1
  Week 3: Extreme Problem | 0
  Week 5: number analyzed (Participants) | 95
  Week 5: No Problem | 43
  Week 5: Slight Problem | 35
  Week 5: Moderate Problem | 16
  Week 5: Severe Problem | 0
  Week 5: Extreme Problem | 1
  Week 7: number analyzed (Participants) | 85
  Week 7: No Problem | 45
  Week 7: Slight Problem | 30
  Week 7: Moderate Problem | 7
  Week 7: Severe Problem | 2
  Week 7: Extreme Problem | 1
  Week 9: number analyzed (Participants) | 90
  Week 9: No Problem | 49
  Week 9: Slight Problem | 27
  Week 9: Moderate Problem | 12
  Week 9: Severe Problem | 1
  Week 9: Extreme Problem | 1
  Week 13: number analyzed (Participants) | 73
  Week 13: No Problem | 40
  Week 13: Slight Problem | 23
  Week 13: Moderate Problem | 6
  Week 13: Severe Problem | 2
  Week 13: Extreme Problem | 2
  Week 17: number analyzed (Participants) | 74
  Week 17: No Problem | 40
  Week 17: Slight Problem | 21
  Week 17: Moderate Problem | 12
  Week 17: Severe Problem | 0
  Week 17: Extreme Problem | 1
  Week 21: number analyzed (Participants) | 63
  Week 21: No Problem | 41
  Week 21: Slight Problem | 15
  Week 21: Moderate Problem | 7
  Week 21: Severe Problem | 0
  Week 21: Extreme Problem | 0
  Week 25: number analyzed (Participants) | 59
  Week 25: No Problem | 29
  Week 25: Slight Problem | 24
  Week 25: Moderate Problem | 4
  Week 25: Severe Problem | 2
  Week 25: Extreme Problem | 0
  Week 37: number analyzed (Participants) | 37
  Week 37: No Problem | 20
  Week 37: Slight Problem | 14
  Week 37: Moderate Problem | 3
  Week 37: Severe Problem | 0
  Week 37: Extreme Problem | 0
  Week 49: number analyzed (Participants) | 23
  Week 49: No Problem | 12
  Week 49: Slight Problem | 9
  Week 49: Moderate Problem | 2
  Week 49: Severe Problem | 0
  Week 49: Extreme Problem | 0
  Week 61: number analyzed (Participants) | 16
  Week 61: No Problem | 8
  Week 61: Slight Problem | 8
  Week 61: Moderate Problem | 0
  Week 61: Severe Problem | 0
  Week 61: Extreme Problem | 0
  Week 73: number analyzed (Participants) | 8
  Week 73: No Problem | 4
  Week 73: Slight Problem | 3
  Week 73: Moderate Problem | 1
  Week 73: Severe Problem | 0
  Week 73: Extreme Problem | 0
  Week 85: number analyzed (Participants) | 4
  Week 85: No Problem | 2
  Week 85: Slight Problem | 2
  Week 85: Moderate Problem | 0
  Week 85: Severe Problem | 0
  Week 85: Extreme Problem | 0
  Week 97: number analyzed (Participants) | 1
  Week 97: No Problem | 1
  Week 97: Slight Problem | 0
  Week 97: Moderate Problem | 0
  Week 97: Severe Problem | 0
  Week 97: Extreme Problem | 0
  Follow-up: number analyzed (Participants) | 30
  Follow-up: No Problem | 16
  Follow-up: Slight Problem | 6
  Follow-up: Moderate Problem | 5
  Follow-up: Severe Problem | 3
  Follow-up: Extreme Problem | 0

25. Secondary Outcome: Pre-dose Plasma Concentration (Ctrough) of Talazoparib
Description: Ctrough was defined as pre-dose plasma concentration during dosing and observed directly from data.
Time Frame: Pre-dose at Week 1, 5, 9 and 13
Population: Pharmacokinetic (PK) population included all participants from the safety population who had at least 1 reportable drug concentration data point. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "Number Analyzed" signifies participants evaluable at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | Talazoparib
Number analyzed (Participants) | 92
nanograms per milliliter
  At Week 1 | 2631.898 (23.2043)
  At Week 5: number analyzed (Participants) | 82
  At Week 5 | 4748.147 (63.2488)
  At Week 9: number analyzed (Participants) | 71
  At Week 9 | 4213.250 (52.8028)
  At Week 13: number analyzed (Participants) | 55
  At Week 13 | 4378.123 (47.5360)

26. Secondary Outcome: Post-dose Plasma Concentration (Ctrough) of Talazoparib
Description: Plasma concentration was measured 2 hours after dosing and observed directly from data.
Time Frame: 2 hours post-dose at Week 1 and 5
Population: PK population included all participants from the safety population who had at least 1 reportable drug concentration data point. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "Number Analyzed" signifies participants evaluable at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | Talazoparib
Number analyzed (Participants) | 31
nanograms per milliliter
  At week 1: number analyzed (Participants) | 25
  At week 1 | 2289.540 (51.0724)
  At Week 5 | 10713.918 (49.4248)

ADVERSE EVENTS:
Time Frame: SAEs and Non-SAEs: Baseline up to 28 days after last dose of study drug (maximum up to 37 months); All-cause mortality: During study included safety follow up and beyond that (approximately 69 months of study)
Description: Same event may appear as both an AE and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Safety population set was analyzed.
Arm/Group | Talazoparib
All-Cause Mortality (participants affected / at risk) | 111/127
Serious Adverse Events (participants affected / at risk) | 51/127
Other Adverse Events (participants affected / at risk) | 124/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Talazoparib (N=127)
Anaemia (Blood and lymphatic system disorders) | 9
Atrial fibrillation (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Disease progression (General disorders) | 5
General physical health deterioration (General disorders) | 2
Pain (General disorders) | 2
Pyrexia (General disorders) | 2
Bronchitis (Infections and infestations) | 1
Neutropenic sepsis (Infections and infestations) | 1
Parotitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Pneumonia aspiration (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 4
Fall (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 2
Platelet count decreased (Investigations) | 2
SARS-CoV-2 test positive (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hemianopia (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Penile pain (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 9
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Talazoparib (N=127)
Anaemia (Blood and lymphatic system disorders) | 67
Constipation (Gastrointestinal disorders) | 27
Diarrhoea (Gastrointestinal disorders) | 22
Nausea (Gastrointestinal disorders) | 45
Vomiting (Gastrointestinal disorders) | 16
Asthenia (General disorders) | 32
Chest pain (General disorders) | 9
Fatigue (General disorders) | 28
Oedema peripheral (General disorders) | 23
Pyrexia (General disorders) | 10
Upper respiratory tract infection (Infections and infestations) | 8
Urinary tract infection (Infections and infestations) | 10
Fall (Injury, poisoning and procedural complications) | 9
Alanine aminotransferase increased (Investigations) | 7
Aspartate aminotransferase increased (Investigations) | 8
Lymphocyte count decreased (Investigations) | 11
Neutrophil count decreased (Investigations) | 22
Platelet count decreased (Investigations) | 27
Weight decreased (Investigations) | 7
White blood cell count decreased (Investigations) | 13
Decreased appetite (Metabolism and nutrition disorders) | 38
Arthralgia (Musculoskeletal and connective tissue disorders) | 19
Back pain (Musculoskeletal and connective tissue disorders) | 19
Bone pain (Musculoskeletal and connective tissue disorders) | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13
Dizziness (Nervous system disorders) | 15
Dysgeusia (Nervous system disorders) | 8
Headache (Nervous system disorders) | 9
Paraesthesia (Nervous system disorders) | 8
Insomnia (Psychiatric disorders) | 8
Haematuria (Renal and urinary disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17
Hot flush (Vascular disorders) | 12
Hypertension (Vascular disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT03148795/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/95/NCT03148795/SAP_002.pdf